CLINICAL TRIAL: NCT05685888
Title: Effect of Ursodeoxycholic Acid on Preventing Covid-19 Infection in Patients With Organ Transplantation: A Multicenter Retrospective Study
Brief Title: Effect of Ursodeoxycholic Acid on Preventing Covid-19 Infection in Patients With Organ Transplantation
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hu Liangshuo, Principal Investigator, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XJTU1AF2023LSK-007
Record Dates: First submitted 2023-01-12; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Organ Transplantation; COVID-19
Keywords: Ursodeoxycholic Acid; COVID-19; Organ transplantation; Immunosuppression
MeSH Terms: conditions — COVID-19 | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Ursodeoxycholic acid (UDCA) group: The Ursodeoxycholic acid (UDCA) group was defined as individuals who have received regular Ursodeoxycholic acid treatments during the two weeks before diagnosed COVID-19 infection (The frequency and dosage of UDCA were also recorded). Subjects matching the characteristics of this group were screened from the database according to inclusion and exclusion criteria, and characteristics of this group were collected and recorded for subsequent analysis.
  Interventions: Other: Medication history
- The non-Ursodeoxycholic acid (non- UDCA) group: The non-Ursodeoxycholic acid (non- UDCA) group was defined as individuals who didn't received regular Ursodeoxycholic acid treatments during the two weeks before diagnosed as COVID-19 infection. Subjects matching the characteristics of this group were screened from the database according to inclusion and exclusion criteria, and characteristics of this group were collected and recorded for subsequent analysis.
  Interventions: Other: Medication history

INTERVENTIONS:
Other: Medication history — The study was retrospective and did not involve the application of interventions

SUMMARY:
Ursodeoxycholic acid is a clinically approved drug which widely used in patients with chronic liver diseases, especially liver transplantation. In China, the COVID-19 infection is in an epidemic state, and the population is generally susceptible to COVID-19. More attention needs to be paid to the prevalence and severity of people taking immunosuppressants after organ transplantation. Recent cohort studies and experiments based on tissue cells, animals and human beings suggest that ursodeoxycholic acid has the potential ability to prevent the entry of COVID-19 into cells, revealing that Ursodeoxycholic acid may be used to prevent the COVID-19 infection. Based on the medical records of patients( already registered on the management website http://www.cltr.org or www.csrkt.org.cn) who received organ transplantation in the First Affiliated Hospital of Xi'an Jiaotong University and the First Affiliated Hospital of Zhengzhou University, this project intends to collect information and data from patients received organ transplantation, aim to understand the COVID-19 infection and severe condition of organ transplantation patients, also explore whether ursodeoxycholic acid has preventive and therapeutic effects on COVID-19 infection and severity rate in patients. This research provides a theoretical basis for further standardizing the prevention and treatment of COVID-19 in patients received organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; 2. Patients received liver or renal transplantation from 2015 to 2022

Exclusion Criteria:

1.Age < 18 years; 2. Multi-organ transplantation; 3. Patients with incomplete information or loss of follow-up; 4.COVID-19 infection before organ transplantation; 5. Patients hospitalized with rejection or other infection within two weeks before COVID-19 diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent liver or renal transplantation from January 1st, 2015, to December 31st, 2022, were retrospectively identified using the database from national transplantation register website and clinical data from the First Affiliated Hospital of Xi'an Jiaotong University and the First Affiliated Hospital of Zhengzhou University.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
The impact of UDCA on the Infection rate of COVID-19 | From January 1,2022 to December 31,2022
  Effect of UDCA on the prevalence and severity of COVID-19 infection in transplantation patients

SECONDARY OUTCOMES:
The impact of UDCA on the rate of severe illness, hospitalization rate and recovery time of COVID-19 | From January 1,2022 to December 31,2022
Protective effects (The Infection rate of COVID-19) of UDCA (different doses) | From January 1,2022 to December 31,2022
Protective effects (The Infection rate of COVID-19) of UDCA in different cohorts (different ages, different immunosuppressants) | From January 1,2022 to December 31,2022

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, MD PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No
The study was based on database from The First Affiliated Hospital of Xi'an JiaoTong University and The First Affiliated Hospital of Zhengzhou University, researchers did not have access to patients' information nor raw data unless approved by the Ethics Committee of The First Affiliated Hospital of Xi'an Jiao Tong University.